CLINICAL TRIAL: NCT06387160
Title: To Determine the Predictors of Reversibility for Acute-on-Chronic Liver Failure at 6-months-A Prospective Study.
Brief Title: To Determine the Predictors of Reversibility for Acute-on-Chronic Liver Failure at 6-months.
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-ACLF-18
Record Dates: First submitted 2024-03-27; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-03

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACLF: 1. Age - 18-75 years
  2. Patients with ACLF(as per APASL guidelines)
  Interventions: Drug: as per institutional protocol

INTERVENTIONS:
Drug: as per institutional protocol — This is an observational study. Treatment will be given to the patients as per institutional protocol

SUMMARY:
ACLF is defined differently in APASL,EASL and AASLD.APASL talks of reversibility in ACLF as per its definition and constitution of Homogenous population with ACLF.The definition of ACLF as per APASL is an acute hepatic insult manifesting as jaundice (serum bilirubin ≥ 5 mg/dL (85 micromol/L) and coagulopathy (INR ≥ 1.5 or prothrombin activity <40%) complicated within 4 weeks by clinical ascites and/or encephalopathy in a patient with previously diagnosed or undiagnosed chronic liver disease/cirrhosis, and is associated with a high 28-day mortality .From the point of view of intensivists, events in form of organ dysfunction , failure or mortality would cumulatively effect the outcome.Reversibility of ACLF syndrome is a feature of the ACLF defined by the AARC criteria, as nearly all the patients included are after the index presentation.With mitigation of the acute insult and over time, the hepatic reserve improves ,fibrosis regresses and the portal pressure decreases. Further, unlike patients with decompensated cirrhosis and similar to patients with ALF, the reversal of coagulopathy preceded the reversal of jaundice,that is ,median time to reversal of syndrome, i.e jaundice and coagulopathy was 7 (4-30)days versus 19 (7-60)days for jaundice, respectively. The median time for reversal of syndrome, i.e, jaundice and coagulopathy ,was 30 days. Baseline albumin, AARC score and Transient elastography predicted long term reversibility .The disease severity assessment is needed for prognostication and to guide the therapy. Furthermore,the available prediction scores have been validated at baseline,but none has been evaluated in a dynamic manner for prognostication in ACLF patients.A DYNAMIC Model that could predict the reversibility in ACLF is urgently required.

DETAILED DESCRIPTION:
Hypothesis:Baseline factors could reliably predict reversibility of ACLF, will help in improved clinical outcomes and risk stratifications.

Aim: To identify the predictors based on clinical, biochemical parameters and noninvasive tests to reliably predict reversibility of ACLF at 6 months

Methodology:

Study population:

* Age - 18-75 years
* Patients with ACLF(as per APASL guidelines) Study design:Prospective Cohort study done at Department of Hepatology,Institute of Liver and Biliary Sciences,New Delhi,India. The study will be conducted in Department of Hepatology .

Duration:2 year Sample size: Assuming that the expected reversibility of ACLF of 60% and desired confidence interval (CI) of 95%,alpha-5% and precision-5%,we need to enroll 370 cases. Considering 28-day mortality rate of around 30% in ACLF patients, we intend to prospectively enroll around 480 patients during the study period.

Monitoring and assessment All patients of ACLF, with acute insult as mentioned in our inclusion criteria, will be prospectively enrolled. Patients will receive standard of care for ACLF. During hospitalization, patients will undergo investigations as per institutional protocol and will receive standard of care as per there acute insult.

Once discharged, all patients will be managed in out-patients as mentioned in the study timeline (figure 1) and will undergo investigations as per the need for monitoring purpose. The list of investigations are mentioned in the figure 2 and is the usual institutional standard of care for medical management of ACLF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age - 18-75 years
2. Patients with ACLF(as per APASL guidelines) admitted in department of Hepatology.
3. Acute Insult-Alcohol,HBV,Auto-immune hepatitis,Viral hepatitis,Drug Induced Liver Injury

Exclusion Criteria:

1. Acute decompensation
2. Complete portal vein thrombosis
3. Hepatocellular carcinoma
4. Tumoral portal vein thrombosis
5. Chronic kidney disease
6. Pregnancy
7. Failure to give consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Age - 18-75 years
  2. Patients with ACLF(as per APASL guidelines)
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
To determine predictors of Reversibility[ Serum Bilirubin < 5mg/dl and PTINR <1.5] at 6 months in Patients of Acute on chronic liver failure as defined by Asian pacific association of study of liver disease[APASL] | 6 months

SECONDARY OUTCOMES:
Change in Asian Pacific Association of Research consortium [AARC] Score from baseline to 90 days and 6 month follow up | 3 and 6 months
Change in liver stiffness measurement [LSM] by Velocity controlled transient elastography[VCTE] at Baseline and 28 Days with values at 90 Days and 6 months. | 28 days, 90-day and 6-months
Change in Spleen stiffness measurement [SSM] by Velocity controlled transient elastography[VCTE] at Baseline and 28 Days with values at 90 Days and 6 months | 28 days, 90-day and 6-months
Change in Grade of fibrosis at Baseline [Day 0 to 28 Day of presentation] measured by Magnetic resonance elastography with 90 Days and 6months values | 3 and 6 months
Proportion of Acute on Chronic Liver failure patients achieving reversibility [Sr Bilirubin <5mg/dl and INR <1.5] as per Asian pacific association of study of liver disease[APASL] at 90 Days. | 3 months
Proportion of Acute on Chronic Liver failure patients achieving reversibility [Sr Bilirubin <5mg/dl and INR <1.5] as per Asian pacific association of study of liver disease[APASL] at 6months. | 6 months
Proportion of Acute on Chronic Liver failure patients maintaining reversibility [Sr Bilirubin <5mg/dl and INR <1.5] as per Asian pacific association of study of liver disease[APASL] at 1year. | 1 year
Proportion of Cirrhotic patients of Acute on Chronic Liver failure patients achieving re compensation at 1year. | 1 year
Proportion of Cirrhotic patients of Acute on Chronic Liver failure patients achieving survival at 1year. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided